CLINICAL TRIAL: NCT02827032
Title: Controlling and Lowering Blood Pressure With the MobiusHD™ - Defining Efficacy Markers
Brief Title: Controlling and Lowering Blood Pressure With the MobiusHD™
Acronym: CALM-DIEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD0328
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MobiusHD™ (Experimental): The MobiusHD device is a self-expanding nitinol implant that is delivered intravascularly to the internal carotid sinus via the delivery catheter.
  Interventions: Device: MobiusHD™

INTERVENTIONS:
Device: MobiusHD™ — The MobiusHD device is a self-expanding nitinol implant that is delivered intravascularly to the internal carotid sinus via the delivery catheter.

SUMMARY:
To perform post-market surveillance and evaluate the performance of the MobiusHD System in subjects with primary resistant hypertension.

DETAILED DESCRIPTION:
The CALM-DIEM Trial is an open-label, prospective, multicenter study for patients who have been selected for treatment with the MobiusHD.

ELIGIBILITY:
Inclusion Criteria:

* Mean 24-hour systolic ABPM is ≥130 mmHg following at least 30 days on a stable antihypertensive medication regimen (no changes in medication or dose), and no more than 28 days prior to implantation.

Exclusion Criteria:

* Known or clinically suspected baroreflex failure or autonomic neuropathy

Substudy Eligibility Criteria: A maximum of 16 patients will be enrolled in the sub-study at one site (Universitair Medisch Centrum Utrecht)

Inclusion Criteria:

- Patients must be eligible for the main study and must have passed all CALM-DIEM study inclusion and exclusion criteria at time of screening

Exclusion Criteria:

* Use of anti-hypertensive drugs directly acting on the sympathetic nervous system that cannot be discontinued safely
* Underlying conditions that prohibit microneurography, performance of a Valsalva maneuver and/or magnetic resonance imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of 24-hour systolic Ambulatory Blood Pressure Measurement (ABPM) | Baseline to ninety (90) days post treatment
  Change in the mean 24-hours systolic Ambulatory Blood Pressure

SECONDARY OUTCOMES:
Incidence of Adverse Events | Baseline to three (3) years post treatment
  Incidence of SAEs and UADEs reported from implantation through three years post treatment

OTHER OUTCOMES:
Substudy Outcome Measure - Change in sympathetic activity | Baseline to 90 days post treatment
  Change in muscle sympathetic nerve activity (burst frequency [bursts/min] and burst incidence [burst/100 heartbeats]) measured by microneurography, from baseline to 90 days post treatment
Substudy Outcome Measure - Change in sympathetic activity | Baseline to 90 days post treatment
  Change in Blood Oxygen Level Dependent (BOLD) activity of central sympathetic nerve circuits (connectivity of the salience network) measured by resting state BOLD fMRI
Substudy Outcome Measure - Change in sympathetic activity | Baseline to 90 days post treatment
  Change in Blood Oxygen Level Dependent (BOLD) activity of central sympathetic nerve circuits (brain(stem) response during the Valsalva maneuver) measured by task-based BOLD fMRI
Substudy Outcome Measure - Change in baroreflex sensitivity | Baseline to 90 days post treatment
  Change sympathetic baroreflex sensitivity (change in muscle sympathetic nerve activity per mmHg blood pressure change) during spontaneous blood pressure fluctuations
Substudy Outcome Measure - Change in baroreflex sensitivity | Baseline to 90 days post treatment
  Change in sympathetic baroreflex sensitivity (change in muscle sympathetic nerve activity per mmHg blood pressure change) during blood pressure changes evoked by the Valsalva maneuver
Substudy Outcome Measure - Change in baroreflex sensitivity | Baseline to 90 days post treatment
  Change in cardiac baroreflex sensitivity (change in heartbeat interval per mmHg blood pressure change) during spontaneous blood pressure fluctuations
Substudy Outcome Measure - Change in baroreflex sensitivity | Baseline to 90 days post treatment
  Change in cardiac baroreflex sensitivity (change in heartbeat interval per mmHg blood pressure change) during blood pressure changes evoked by the Valsalva maneuver

CONTACTS AND LOCATIONS:
Locations (22):
- Germany (9):
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - CVC Frankfurt, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Charite Berlin, Berlin
  - Asklepiod Klinik Hamburg, Hamburg
  - Universitatsklinikum des Saarlandes, Homburg
- Netherlands (6):
  - HagaZiekenhuis, The Hague, AA
  - St. Antonius Ziekenhuis, Nieuwegein, EM
  - Maastricht UMC+, Maastricht, HX
  - Radboud University Medical Center, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Isala, Zwolle
- United Kingdom (7):
  - Queen Elizabeth University Hospital - Glasgo, Glasgow, Scotland
  - Golden Jubilee National Hospital, Glasgow, Scotland
  - The Royal Sussex County Hospital, Brighton
  - St. Bartholomew's Hospital, London
  - St. Thomas' Hospital, London
  - University College London Hospital, London
  - Manchester University, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Groenland EH, van Kleef MEAM, Hendrikse J, Spiering W, Siero JCW. The effect of endovascular baroreflex amplification on central sympathetic nerve circuits and cerebral blood flow in patients with resistant hypertension: A functional MRI study. Front Neuroimaging. 2022 Jul 25;1:924724. doi: 10.3389/fnimg.2022.924724. eCollection 2022. PMID 37555165
- [Derived] van Kleef MEAM, Heusser K, Diedrich A, Oey PL, Tank J, Jordan J, Blankestijn PJ, Williams B, Spiering W. Endovascular baroreflex amplification and the effect on sympathetic nerve activity in patients with resistant hypertension: A proof-of-principle study. PLoS One. 2021 Nov 16;16(11):e0259826. doi: 10.1371/journal.pone.0259826. eCollection 2021. PMID 34784359